CLINICAL TRIAL: NCT01175876
Title: The Effect Of Remote Limb Ischemic Preconditioning For Carotid Artery Stenting
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Xunming Ji, XuanWu Hospital，Capital medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIPC2010
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Stroke; TIA; Coronary Stenosis
Keywords: MMSE; NSE; S100B; hsCRP; DWI-MRI
MeSH Terms: conditions — Stroke; Coronary Stenosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Device: RIPC RIPC consisted of five 5-min cycles of right upper arm ischemia/reperfusion, which was induced by an automated cuff-inflator placed on the right upper arm which was inflated to 200 mmHg for 5mins followed by deflating the cuff for 5mins Procedure: Carotid Artery Stenting
  Interventions: Device: remote limb ischemic preconditioning; Procedure: Carotid Artery Stenting
- 2 (Sham Comparator): Procedure: Carotid Artery Stenting
  Interventions: Procedure: Carotid Artery Stenting

INTERVENTIONS:
Device: remote limb ischemic preconditioning — Remote limb ischemic preconditioning consisted of five 5-min cycles of right upper arm ischemia/reperfusion, which was induced by an automated cuff-inflator placed on the right upper arm which was inflated to 200 mmHg for 5mins followed by deflating the cuff for 5mins
  Arms: 1
Procedure: Carotid Artery Stenting — Carotid Artery Stenting is an invasive therapy of carotid stenosis.

SUMMARY:
Remote limb ischemic preconditioning is neuro-protective and anti-inflammatory for ischemia- reperfusion injury. As the extent of its effect is unknown, the investigators will use clinical outcome, serum biochemical markers and diffusion-weighted magnetic resonance imaging (DW-MRI)to determine the extent of its neuro-protective and anti-inflammatory effect.

DETAILED DESCRIPTION:
BACKGROUND: Brain ischemia and injury contributed to perioperative morbidity and mortality in Carotid Artery Stenting. Remote ischemic preconditioning (RIPC) is a phenomenon whereby brief periods of ischemia followed by reperfusion in one organ provide systemic protection from prolonged ischemia. To investigate whether remote preconditioning protects the brain injury in patients undergoing elective Carotid Artery Stenting, a randomized trial will be performed in current study.

DESIGNING 60 patients will be randomized to Carotid Artery Stenting with RIPC group or conventional Carotid Artery Stenting group (control). RIPC consisted of five 5-min cycles of right upper arm ischemia/reperfusion, which was induced by an automated cuff-inflator placed on the right upper arm which was inflated to 200 mmHg for 5mins followed by deflating the cuff for 5mins. Cerebral injury was assessed by S-100b, NSE, hs-CRP and MMSE test in different time points.

ELIGIBILITY:
Inclusion Criteria:Patients referred for elective Carotid Artery Stenting were participate in the study at the time of scheduling for operation.

1. Symptomatic patient, as evidenced by transient ischemic attack (TIA), amaurosis fugax, minor or non-disabling stroke(in the hemisphere supplied by the target vessel), within 180 days of the randomization date.
2. Discrete lesion located in the internal carotid artery(ICA), and the degree of carotid stenosis ≥50% defined as:

   Stenosis ≥70% by ultrasound. Stenosis ≥50% by angiography (based on NASCET Criteria)
3. Appropriate for carotid stenting. Candidates for Carotid Artery Stenting meet all other inclusion requirements.

Exclusion Criteria:

1. Evolving stroke
2. Untoward reaction to anesthesia
3. Intolerance or allergic reaction to associated medications, including aspirin(ASA) and clopidogrel.
4. Prior major ipsilateral stroke that may confound study endpoints.
5. Severe dementia.
6. Hemorrhagic transformation of an ischemic stroke within the past 60 days.
7. Chronic atrial fibrillation.
8. MI within previous 30 days.
9. High risk surgical candidate defined as the CREST test.
10. Bilateral upper limb arteries are severe stenotic or occlusion.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
cognitive disorder assessment | 2 days
  1.The Mini-Mental State Examination( MMSE) test: The difference in MMSE score among patients treated with preconditioning and those not treated.
serum biomarkers | 2 days
  Serum biomarkers of brain injury and flammatory: The difference in NSE, S-100b and hs-CRP level among patients treated with preconditioning and those not treated.
new brain lesions | 2DAYS
  The new lesions at DWI-MRI within postoperation 48 hours: The difference in new lesions in the DWI-MRI 48 hours postoperatively among patients treated with preconditioning and those not treated.

SECONDARY OUTCOMES:
composite endpoint of any stroke,MI,or death | 3months
  The composite endpoint of any stroke ,MI, or death at 30-day and 90-day after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, M.D.,Ph.D., Study Chair — Proffessor
Locations (1):
- Yumin Luo, Beijing, Beijing Municipality, China